CLINICAL TRIAL: NCT03492983
Title: Effect of High Cocoa Content Chocolate on Vascular Function, Body Composition, Health-related Quality of Life and Cognitive Performance in Postmenopausal Women.
Brief Title: Effect of High Cocoa Content Chocolate on Health in Postmenopausal Women.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion y Formacion en Ciencias de la Salud (Other)
Collaborators: Castilla-León Health Service (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: GRS 1583/B/17
Record Dates: First submitted 2018-03-23; First posted 2018-04-10 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Postmenopausal Women
Keywords: Cocoa; Vascular function; Body composition; Quality of life; Cognitive performance; Postmenopausal women

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): No intervention
- Intervention group (Experimental): Addition of 10 g/day of high cocoa content chocolate to the usual diet for six months
  Interventions: Dietary Supplement: Intervention group

INTERVENTIONS:
Dietary Supplement: Intervention group — 10 g/day of high cocoa content chocolate for six months.
  Arms: Intervention group

SUMMARY:
This is a randomized clinical trial aimed at postmenopausal women aged 50 to 64 years old selected in urban primary care centers of two centers (Spain). Its objective is to evaluate the effects of the additional intake of high cocoa content chocolate on blood pressure, vascular function, body composition, quality of life and cognitive performance.

DETAILED DESCRIPTION:
* Objective: To assess the effect at 6 months of the additional intake of 10 g/day of high cocoa content chocolate for 6 months on blood pressure, vascular function, body composition, quality of life and cognitive performance in postmenopausal women.
* Design and setting: A randomized clinical trial of two parallel groups. Population: 140 postmenopausal women, 50 to 64 aged will be included, selected by consecutive sampling in two primary care centers.
* Measurements and intervention: Vascular function (blood pressure, augmentation index and Cardio-Ankle Vascular Index), body composition and health-related quality of life will be evaluated. The intervention group will receive a daily supplement of high cocoa content chocolate for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Women in postmenopausal period defined as 12 consecutive months of amenorrhea.

Exclusion Criteria:

* Older than 65 years.
* Cardiovascular disease (acute myocardial infarction, stroke).
* Arterial hypertension on treatment.
* Diabetes mellitus.
* Dyslipidemia (total cholesterol >250 mg/dL or in lipid-lowering therapy).
* Clinically demonstrable neurological and/or neuropsychological disorders.
* Hormone replacement therapy.
* Allergy and/or intolerance to cocoa or any of the components of the supplement.
* Hypocaloric diet.
* Any other circumstance that the investigators consider could interfere with the study procedures.

Ages: 50 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 6 months
  Measurement by oscillometric method (mmHg)

SECONDARY OUTCOMES:
Arterial stiffness | 6 months
  Measurement by Brachial-ankle pulse wave velocity (m/s)
Wave reflection | 6 months
  Measurement by central and peripheral augmentation index
Body composition | 6 months
  Measurement by body fat percentage
Quality of life | 6 months
  Measurement by Cervantes Scale (Score between 0 (poor quality) and 155 (high quality)
Cognitive performance | 6 months
  Measurement by executive function

CONTACTS AND LOCATIONS:
Overall Officials: Jose I Recio-Rodriguez, PhD, Principal Investigator — University of Salamanca
Locations (1):
- Instituto Biosanitario de Salamanca. Research unit La Alamedilla, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garcia-Yu IA, Garcia-Ortiz L, Gomez-Marcos MA, Rodriguez-Sanchez E, Mora-Simon S, Maderuelo-Fernandez JA, Recio-Rodriguez JI. Effects of cocoa-rich chocolate on cognitive performance in postmenopausal women. A randomised clinical trial. Nutr Neurosci. 2022 Jun;25(6):1147-1158. doi: 10.1080/1028415X.2020.1840119. Epub 2020 Nov 15. PMID 33190575
- [Derived] Garcia-Yu IA, Garcia-Ortiz L, Gomez-Marcos MA, Alonso-Dominguez R, Gonzalez-Sanchez J, Mora-Simon S, Gonzalez-Manzano S, Rodriguez-Sanchez E, Maderuelo-Fernandez JA, Recio-Rodriguez JI. Vascular and cognitive effects of cocoa-rich chocolate in postmenopausal women: a study protocol for a randomised clinical trial. BMJ Open. 2018 Dec 14;8(12):e024095. doi: 10.1136/bmjopen-2018-024095. PMID 30552275